CLINICAL TRIAL: NCT02118168
Title: OBSERVATIONAL STUDY FOR THE EXTENDED FOLLOW-UP OF THE PATIENTS ENROLLED IN THE PHASE II THERAPEUTIC CLINICAL TRIAL ISS T-002
Brief Title: Observational Study for the Extended Follow-up of the Patients Enrolled in the Therapeutic Clinical Trial ISS T-002
Acronym: ISST-002 EF-UP
Status: Completed | Type: Observational
Sponsor: Barbara Ensoli, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Barbara Ensoli, MD, PhD, PhD, Istituto Superiore di Sanità
Organization: Istituto Superiore di Sanità (Other)
Other Study IDs: ISS T-002 EF-UP
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: HIV Infection
Keywords: HIV; HAART; Tat Protein
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: All patients that participated to the therapeutic phase II trial of the Tat vaccine "ISS T-002" and that received at least 3 immunizations and reached 48-weeks of follow-up.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention is foreseen in this Observational Study

SUMMARY:
An observational study to prospectively follow-up the patients enrolled in the ISS T-002 clinical trial up to 132 weeks. The primary endpoint of this study is to evaluate the persistence, in term of frequency, magnitude and quality, of the anti-Tat humoral and cellular immune response in the HIV-1 infected individuals who participated to the ISS T-002 and who have received at least 3 immunizations. The secondary endpoint is to define and validate novel laboratory tests for future efficacy clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in the ISS T-002 trial, having received at least 3 immunizations;
* A follow-up of at least 48 weeks during the ISS T-002 study;
* Availability to participate in the extended follow-up study;
* Signed informed consent.

Exclusion Criteria:

* The absence of any of the above criteria will exclude the subjects from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HAART-treated patients who participated to the therapeutic phase II trial of the Tat vaccine "ISS T-002" and received at least 3 immunizations and reached 48-weeks of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
anti-Tat humoral immune response | Every 3 months, up to 2.5 years
  The primary endpoint of the study is to evaluate the persistence, in term of frequency, magnitude, and quality of the anti-Tat humoral immune response in HAART-treated patients previously immunize with Tat in the ISS T-002 phase II clinical trial.

SECONDARY OUTCOMES:
Testing of the additional Immunological parameters detailed below as a second line testing | Every 3 months, up to 2.5 years
  The secondary endpoint of the study is to identify and validate immunological testing for future efficacy vaccine clinical trials, as follows: Lymphoproliferative response to Tat, anti-Tat γIFN, IL4 and IL2 production; In vitro neutralization of Tat activity (Tat/Env uptake); Lymphocyte subsets; Anti-Tat IgG subclasses; Epitope mapping of anti-Tat IgM and IgG; Anti-HIV regulatory and structural proteins antibodies; ADCC; Neutralization of Tat activity by rescue assay; Neutralization of primary HIV isolates; Anti-CCR5 and Anti-CD4 antibodies; Lymphoproliferative response to Env, mitogens and recall antigens In vitro γIFN, IL4 and IL2 production in response to Tat (ICS) and to Env (ICS/Elispot); B cells phenotype; Characterization of Treg cells; PBMC ICS for granzyme, perforin, cytokines and chemokines; Th1 and Th2 cytokines and chemokines; Lymphocytes spontaneous cell death; B cell cloning; Characterization of clono-specific antibodies; Serum/plasma determination of sCD4.
Testing of virological parameters detailed below, as a second line testing | Every 3 months, up to 2.5 years
  The secondary endpoint of the study is to identify and validate virological testing for future efficacy vaccine clinical trials, as follows: HIV-1 plasma viremia (viral RNA copies), HIV-1 sequencing and virus phylogenetic analysis, Genotypic resistance, Viral tropism, Anti-HBV antibodies, HBV antigens (HbsAg, HbeAg), Anti-HCV antibodies and plasma viremia, HHV-8 antibodies and plasma viremia, HIV-1 Proviral DNA copies.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ensoli, MD, PHD, Study Director — Istituto Superiore di Sanità
Locations (8):
- Italy (8):
  - Divisione di Malattie Infettive Azienda Ospedaliera S. Gerardo, Monza, MB
  - Divisione Malattie Infettive - AO Ospedale Policlinico Consorziale, Bari
  - Ambulatorio Malattie Infettive - AO Universitaria, Ferrara
  - Unità Operativa di Malattie Infettive - Ospedale S.M. Annunziata, Florence
  - U. O. di Malattie Infettive Centro di Ricerca e Cura Patologie HIV correlate - Ospedale San Raffaele, Milan
  - Istituto di Malattie Infettive e Tropicali - AO Luigi Sacco, Milan
  - Divisione di Malattie Infettive - AO Universitaria Policlinico, Modena
  - U.O.C. Dermatologia Infettiva ed Allergologica - IFO San Gallicano, Roma

REFERENCES:
- [Background] Longo O, Tripiciano A, Fiorelli V, Bellino S, Scoglio A, Collacchi B, Alvarez MJ, Francavilla V, Arancio A, Paniccia G, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Phase I therapeutic trial of the HIV-1 Tat protein and long term follow-up. Vaccine. 2009 May 26;27(25-26):3306-12. doi: 10.1016/j.vaccine.2009.01.090. Epub 2009 Feb 7. PMID 19208456
- [Background] Bellino S, Francavilla V, Longo O, Tripiciano A, Paniccia G, Arancio A, Fiorelli V, Scoglio A, Collacchi B, Campagna M, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Parallel conduction of the phase I preventive and therapeutic trials based on the Tat vaccine candidate. Rev Recent Clin Trials. 2009 Sep;4(3):195-204. doi: 10.2174/157488709789957529. PMID 20028332
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Tripiciano A, Longo O, Bellino S, Francavilla V, Paniccia G, Arancio A, Scoglio A, Collacchi B, Ruiz Alvarez MJ, Tambussi G, Tassan Din C, Palamara G, Latini A, Antinori A, D'Offizi G, Giuliani M, Giulianelli M, Carta M, Monini P, Magnani M, Garaci E. The preventive phase I trial with the HIV-1 Tat-based vaccine. Vaccine. 2009 Dec 11;28(2):371-8. doi: 10.1016/j.vaccine.2009.10.038. Epub 2009 Oct 29. PMID 19879233
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Monini P, Magnani M, Garaci E. The therapeutic phase I trial of the recombinant native HIV-1 Tat protein. AIDS. 2008 Oct 18;22(16):2207-9. doi: 10.1097/QAD.0b013e32831392d4. PMID 18832884
- [Background] Ensoli B, Bellino S, Tripiciano A, Longo O, Francavilla V, Marcotullio S, Cafaro A, Picconi O, Paniccia G, Scoglio A, Arancio A, Ariola C, Ruiz Alvarez MJ, Campagna M, Scaramuzzi D, Iori C, Esposito R, Mussini C, Ghinelli F, Sighinolfi L, Palamara G, Latini A, Angarano G, Ladisa N, Soscia F, Mercurio VS, Lazzarin A, Tambussi G, Visintini R, Mazzotta F, Di Pietro M, Galli M, Rusconi S, Carosi G, Torti C, Di Perri G, Bonora S, Ensoli F, Garaci E. Therapeutic immunization with HIV-1 Tat reduces immune activation and loss of regulatory T-cells and improves immune function in subjects on HAART. PLoS One. 2010 Nov 11;5(11):e13540. doi: 10.1371/journal.pone.0013540. PMID 21085635
- [Background] Monini P, Cafaro A, Srivastava IK, Moretti S, Sharma VA, Andreini C, Chiozzini C, Ferrantelli F, Cossut MR, Tripiciano A, Nappi F, Longo O, Bellino S, Picconi O, Fanales-Belasio E, Borsetti A, Toschi E, Schiavoni I, Bacigalupo I, Kan E, Sernicola L, Maggiorella MT, Montin K, Porcu M, Leone P, Leone P, Collacchi B, Palladino C, Ridolfi B, Falchi M, Macchia I, Ulmer JB, Butto S, Sgadari C, Magnani M, Federico MP, Titti F, Banci L, Dallocchio F, Rappuoli R, Ensoli F, Barnett SW, Garaci E, Ensoli B. HIV-1 tat promotes integrin-mediated HIV transmission to dendritic cells by binding Env spikes and competes neutralization by anti-HIV antibodies. PLoS One. 2012;7(11):e48781. doi: 10.1371/journal.pone.0048781. Epub 2012 Nov 13. PMID 23152803
- [Background] Ensoli B, Fiorelli V, Ensoli F, Cafaro A, Titti F, Butto S, Monini P, Magnani M, Caputo A, Garaci E. Candidate HIV-1 Tat vaccine development: from basic science to clinical trials. AIDS. 2006 Nov 28;20(18):2245-61. doi: 10.1097/QAD.0b013e3280112cd1. No abstract available. PMID 17117011
- [Background] Butto S, Fiorelli V, Tripiciano A, Ruiz-Alvarez MJ, Scoglio A, Ensoli F, Ciccozzi M, Collacchi B, Sabbatucci M, Cafaro A, Guzman CA, Borsetti A, Caputo A, Vardas E, Colvin M, Lukwiya M, Rezza G, Ensoli B; Tat Multicentric Study Group. Sequence conservation and antibody cross-recognition of clade B human immunodeficiency virus (HIV) type 1 Tat protein in HIV-1-infected Italians, Ugandans, and South Africans. J Infect Dis. 2003 Oct 15;188(8):1171-80. doi: 10.1086/378412. Epub 2003 Sep 30. PMID 14551888
- [Background] Rezza G, Fiorelli V, Dorrucci M, Ciccozzi M, Tripiciano A, Scoglio A, Collacchi B, Ruiz-Alvarez M, Giannetto C, Caputo A, Tomasoni L, Castelli F, Sciandra M, Sinicco A, Ensoli F, Butto S, Ensoli B. The presence of anti-Tat antibodies is predictive of long-term nonprogression to AIDS or severe immunodeficiency: findings in a cohort of HIV-1 seroconverters. J Infect Dis. 2005 Apr 15;191(8):1321-4. doi: 10.1086/428909. Epub 2005 Mar 14. PMID 15776379
- [Background] Cafaro A, Caputo A, Maggiorella MT, Baroncelli S, Fracasso C, Pace M, Borsetti A, Sernicola L, Negri DR, Ten Haaft P, Betti M, Michelini Z, Macchia I, Fanales-Belasio E, Belli R, Corrias F, Butto S, Verani P, Titti F, Ensoli B. SHIV89.6P pathogenicity in cynomolgus monkeys and control of viral replication and disease onset by human immunodeficiency virus type 1 Tat vaccine. J Med Primatol. 2000 Aug;29(3-4):193-208. doi: 10.1034/j.1600-0684.2000.290313.x. PMID 11085582
- [Background] Bellino S, Tripiciano A, Picconi O, Francavilla V, Longo O, Sgadari C, Paniccia G, Arancio A, Angarano G, Ladisa N, Lazzarin A, Tambussi G, Nozza S, Torti C, Foca E, Palamara G, Latini A, Sighinolfi L, Mazzotta F, Di Pietro M, Di Perri G, Bonora S, Mercurio VS, Mussini C, Gori A, Galli M, Monini P, Cafaro A, Ensoli F, Ensoli B. The presence of anti-Tat antibodies in HIV-infected individuals is associated with containment of CD4+ T-cell decay and viral load, and with delay of disease progression: results of a 3-year cohort study. Retrovirology. 2014 Jun 24;11:49. doi: 10.1186/1742-4690-11-49. PMID 24961156
- [Background] Ensoli B, Cafaro A, Monini P, Marcotullio S, Ensoli F. Challenges in HIV Vaccine Research for Treatment and Prevention. Front Immunol. 2014 Sep 8;5:417. doi: 10.3389/fimmu.2014.00417. eCollection 2014. PMID 25250026
- [Background] Ensoli F, Cafaro A, Casabianca A, Tripiciano A, Bellino S, Longo O, Francavilla V, Picconi O, Sgadari C, Moretti S, Cossut MR, Arancio A, Orlandi C, Sernicola L, Maggiorella MT, Paniccia G, Mussini C, Lazzarin A, Sighinolfi L, Palamara G, Gori A, Angarano G, Di Pietro M, Galli M, Mercurio VS, Castelli F, Di Perri G, Monini P, Magnani M, Garaci E, Ensoli B. HIV-1 Tat immunization restores immune homeostasis and attacks the HAART-resistant blood HIV DNA: results of a randomized phase II exploratory clinical trial. Retrovirology. 2015 Apr 29;12:33. doi: 10.1186/s12977-015-0151-y. PMID 25924841
- [Background] Cafaro A, Tripiciano A, Sgadari C, Bellino S, Picconi O, Longo O, Francavilla V, Butto S, Titti F, Monini P, Ensoli F, Ensoli B. Development of a novel AIDS vaccine: the HIV-1 transactivator of transcription protein vaccine. Expert Opin Biol Ther. 2015;15 Suppl 1:S13-29. doi: 10.1517/14712598.2015.1021328. Epub 2015 Jun 22. PMID 26096836
- [Derived] Sgadari C, Monini P, Tripiciano A, Picconi O, Casabianca A, Orlandi C, Moretti S, Francavilla V, Arancio A, Paniccia G, Campagna M, Bellino S, Meschiari M, Nozza S, Sighinolfi L, Latini A, Muscatello A, Saracino A, Di Pietro M, Galli M, Cafaro A, Magnani M, Ensoli F, Ensoli B. Continued Decay of HIV Proviral DNA Upon Vaccination With HIV-1 Tat of Subjects on Long-Term ART: An 8-Year Follow-Up Study. Front Immunol. 2019 Feb 13;10:233. doi: 10.3389/fimmu.2019.00233. eCollection 2019. PMID 30815001